CLINICAL TRIAL: NCT03210909
Title: Pharmacokinetics and Metabolism of [14C] BMS-986231 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV013-022
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Heart Decompensation, Acute
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986231 Intravenous Infusion (Experimental): A single continuous intravenous infusion of BMS-986231
  Interventions: Drug: BMS-986231

INTERVENTIONS:
Drug: BMS-986231 — BMS-986231

SUMMARY:
An intravenous infusion in healthy subjects to obtain information about the absorption, metabolism, and excretion (AME) of BMS-986231

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Target population: Healthy males with no clinically significant deviations from normal in medical history, physical examinations, vital signs, electrocardiograms (ECGs), physical measurements, and clinical laboratory tests
* Body weight between 75 and 95 kg, inclusive; body mass index (BMI) between 18 to 32 kg/m2.

Exclusion Criteria:

* History of chronic illness
* Chronic headaches
* Recurrent dizziness
* Personal or family history of heart disease
* Personal history of bleeding diathesis

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time Zero to Time of Last Quantifiable Concentration (AUC[0-T]) | Up to 8 days
  Measured by plasma concentrations
Percent of Total Radioactivity Recovered in All Excreta (% total) | Up to 8 days
  Measured by plasma urine, feces, and vomit (if applicable) volumes and radioactivity counts
Half-Life (T-HALF) | Up to 8 days
  Measured by plasma concentrations
Total Body Clearance (CLT) | Up to 8 days
  Measured by plasma concentrations
Volume of Distribution during Terminal Elimination Phase (Vz/F) | Up to 8 days
  Measured by plasma concentrations
Time to Maximum Observed Concentration (Tmax) | Up to 8 days
  Measured by plasma concentrations

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 8 days
  Measured by investigator assessment
Results of electrocardiogram tests (ECGs) | Up to 8 days
  Measured by investigator assessment
Results of vital sign measurements | Up to 8 days
  Measured by investigator assessment
Results of clinical laboratory tests | Up to 8 days
  Measured by investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx